CLINICAL TRIAL: NCT07172035
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) for Recompensation in Patients With Decompensated Cirrhosis: A Multicenter Prospective Cohort Study
Brief Title: The Impact of Transjugular Intrahepatic Portosystemic Shunt on Recompensation in Patients With Decompensated Liver Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Zhongnan Hospital (Other); Yichang Central People's Hospital (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); Jiangxi Provincial People's Hopital (Other); The Central Hospital of Huanggang (Other); Second Xiangya Hospital of Central South University (Other); Shengjing Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanxi Provincial People's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); The Third Xiangya Hospital of Central South University (Other); Fujian Medical University Union Hospital (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yaowei Bai, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: TIPS-Recompensation
Record Dates: First submitted 2025-09-05; First posted 2025-09-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis; Decompensation; Transjugular Intrahepatic Portosystemic Shunt (TIPS); Survival Analysis
Keywords: Cirrhosis; decompensation; transjugular intrahepatic portosystemic shunt (TIPS); Survival analysis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recompensation group: Refers to the group of patients who simultaneously meet the three core criteria of "etiology cure", "resolution of decompensation events" and "sustained improvement of liver function" at 1 year after TIPS creation
- Non-Recompensation Group: Refers to the group of patients who fail to meet the three core criteria of "etiology cure", "resolution of decompensation events" and "sustained improvement of liver function" at 1 year after TIPS creation.

SUMMARY:
The traditional view holds that the natural course of cirrhosis is a unidirectional process, characterized by irreversible progression from the compensated stage to the decompensated stage, and is highly likely to develop further decompensation events or even death. However, a growing body of evidence suggests that the natural course of cirrhosis is not always unidirectional - after the removal of the etiology, the structural and functional changes of the liver may be partially reversed. This understanding has given rise to the concept of "liver recompensation," which has been standardized at the Baveno VII Consensus Conference. Notably, in a cohort of patients with alcohol-related cirrhosis, 18% achieved recompensation, which was significantly associated with a reduction of more than 90% in liver-related mortality. In patients with hepatitis B-related cirrhosis, 6% achieved recompensation after treatment with nucleos(t)ide analogs, with a similar improvement in mortality.

Transjugular intrahepatic portosystemic shunt (TIPS) is a well-established therapy for complications related to portal hypertension, including gastroesophageal variceal bleeding, refractory ascites, and hepatic hydrothorax. Compared with standard treatment, TIPS has been proven to reduce the incidence of further decompensation and improve transplant-free survival. However, due to portal blood shunting, the risks of abnormal liver function and hepatic encephalopathy (HE) also increase. It is worth noting that TIPS is not included in the definition of recompensation in the Baveno VII Consensus. Therefore, whether patients with cirrhosis who undergo TIPS treatment can achieve recompensation and which factors determine the probability of recompensation remain unknown. More importantly, the impact of recompensation on the risk of HCC development and mortality in TIPS patients has not been studied prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Diagnosed with decompensated liver cirrhosis (diagnostic criteria: positive liver histopathological examination, or comprehensive judgment based on clinical symptoms, biochemical indicators and imaging features);
3. The etiology of liver cirrhosis is intervenable (including hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, alcoholic liver disease (ALD), etc.);
4. Patients with indications for Transjugular Intrahepatic Portosystemic Shunt (TIPS) treatment of cirrhotic portal hypertension, such as those with cirrhotic portal hypertension-related esophagogastric variceal bleeding refractory to endoscopic treatment, and patients with refractory ascites caused by cirrhotic portal hypertension;
5. Obtained informed consent signed by the patient or their family members.

Exclusion Criteria:

1. Compensated liver cirrhosis at the time of TIPS treatment (without decompensated events such as ascites, hepatic encephalopathy, or esophagogastric variceal bleeding);
2. TIPS performed for the treatment of non-cirrhotic portal hypertension (e.g., idiopathic portal hypertension, Budd-Chiari syndrome, sinusoidal obstruction syndrome, etc.);
3. Patients complicated with malignant tumors such as hepatocellular carcinoma (HCC), renal cell carcinoma, or lung cancer prior to TIPS;
4. Patients with severe cardiopulmonary dysfunction or a Model for End-Stage Liver Disease (MELD) score > 18;
5. Pregnant patients;
6. Patients with uncontrolled systemic infection or inflammation;
7. Patients with severe coagulation disorders;
8. Patients allergic to contrast medium.

Criteria for Termination/Withdrawal from the Study:

1. Patients with Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure failure due to various reasons;
2. Patients who voluntarily request to withdraw from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of this research consists of patients with decompensated cirrhotic portal hypertension who meet the predefined inclusion and exclusion criteria and undergo transjugular intrahepatic portosystemic shunt (TIPS) treatment.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
1-year post-TIPS recompensation rate | 1 year
  It refers to the proportion of patients who meet the standardized recompensation criteria (etiology cure, resolution of decompensation events and sustained improvement of liver function) at 12 months after TIPS.

SECONDARY OUTCOMES:
Identification of factors associated with recompensation at 1 year after TIPS | 1 year
  It refers to the screening and confirmation of potential factors that may affect whether patients achieve recompensation at 1 year after TIPS. Cox Univariate analysis and multivariate regression analysis will be used to identify independent factors associated with recompensation, providing a basis for individualized intervention strategies to improve the recompensation rate of TIPS patients.
Impact of recompensation on the risk of hepatocellular carcinoma (HCC) development | 1 year
  It refers to the comparison of the incidence of HCC between the recompensation group and the non-recompensation group during the follow-up period after TIPS surgery.
Impact of recompensation after Transjugular Intrahepatic Portosystemic Shunt on patients' risk of death | 1 year
  At 12 months after Transjugular Intrahepatic Portosystemic Shunt (TIPS), patients were divided into the recompensation group and the non-recompensation group based on whether they met the recompensation criteria, and the Log-rank test was used to analyze the differences in survival outcomes between the two groups.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Second Xiangya Hospital, Central South University, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Fujian Medical University Union Hospital, Fuzhou
  - Huanggang Central Hospital, Huanggang
  - Jingzhou Central Hospital, Jingzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Shengjing Hospital of China Medical University, Shenyang
  - Shanxi Provincial People's Hospital, Taiyuan
  - Renmin Hospital of Wuhan University, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Xiangyang Central Hospital, Xiangyang
  - Yichang Central People's Hospital, Yichang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided